CLINICAL TRIAL: NCT04369898
Title: A Multi-centric Study of the Combined Sensitivity and Specificity of Cortical Lesions and Central Vein Sign for MS Diagnosis and Differential Diagnosis
Brief Title: Combined Sensitivity and Specificity of Cortical Lesions and Central Vein Sign for MS Diagnosis and Differential Diagnosis
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-00765; me20Granziera
Record Dates: First submitted 2020-04-27; First posted 2020-04-30 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Multiple Sclerosis)
Keywords: cortical lesions; leuco-cortical lesions; central vein sign
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Image analysis/ Central vein detection — Image analysis/ Central vein detection will be performed using a fully automated approach based on an ensemble of 3D convolutional neural Networks. The method is applied to T1w, T2w and T2*w data . Results will be manually reviewed by 2 experts in CVs detection. MRI data must have been collected at 3 Tesla (3T) between 1990 and 2020 and must include T1 w, T2 w, T2-star based sequence (CVs detection).
Other: Image analysis/ Automatic cortical lesion detection — Image analysis/ Automatic cortical lesion detection will be performed by using a convolutional neural network-based method. MRI data must have been collected at 3T between 1990 and 2020 and must include Double inversion recovery (DIR)/Phase-Sensitive Inversion Recovery (PSIR)/Magnetization Prepared - 2- RApid Gradient Echo Gradient Echo (MP2RAGE) (eventually also high spatial resolution Magnetization Prepared - RApid Gradient Echo (MPRAGE)) for cortical lesion detection.

SUMMARY:
This study investigates the specificity/sensitivity of the combined presence of cortical lesions (CLs)/leuco-cortical lesions (LCLs) and central veins sign (CVs) for multiple sclerosis (MS) diagnosis and differential diagnosis.

DETAILED DESCRIPTION:
CLs and LCLs may be detected at 3 Tesla (T) MRI by using dedicated sequences. 3D Double inversion recovery (DIR), Phase-Sensitive Inversion Recovery (PSIR), Magnetization Prepared - RApid Gradient Echo (MPRAGE) and Magnetization Prepared - 2- RApid Gradient Echo (MP2RAGE) have all shown variable sensitivity to CLs and LCLs. The central vein sign (CVS, i.e. the detection of a central vessel in a focal lesion) has been recently proposed as a biomarker for distinguishing between MS and not and not MS. Both the presence of CL and CVs brings high sensitivity and specificity in distinguishing MS from not MS patients; whether their combination achieves higher sensitivity and specificity to MS diagnosis and differential diagnosis is to date not know. This study investigates the specificity/sensitivity of the combined presence of cortical lesions (CLs)/leuco-cortical lesions (LCLs) and central veins sign (CVs) for multiple sclerosis (MS) diagnosis and differential diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and MRI data of patients with MS or MS mimics (migraine, vasculitis, diabetes, neuromyelitis optica spectrum disorder)
* MRI data must have been collected at 3T between 1990 and 2020 and must include T1 w, T2 w, T2-star based sequence (CVs detection) and DIR/PSIR/MP2RAGE (eventually also high spatial resolution MPRAGE) for cortical lesion detection

Exclusion Criteria:

* Unavailability of institutional informed consent
* Unclear diagnosis
* Other neurological or psychiatric diseases.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: MRI and clinical coded data will be collected from some of the European centers that belong to the MAGNIMS consortium (Oxord University, University College London, University Hospital Vall d'Hebron (Barcelona), Verona University) as well as from Basel University hospital. MAGNIMS members and associate centers have a common data-sharing agreement (enclosed).
  MAGNIMS is an independent European network of academics that share a common interest in the study of multiple sclerosis (MS) using magnetic resonance imaging (MRI). MRI data must have been collected at 3T between 1990 and 2020.
Sampling Method: Probability Sample
Enrollment: 1051 (Actual)
Dates: Start 2010-06-01 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2023-09 (Actual)

PRIMARY OUTCOMES:
differentiation between patients with MS and clinically isolated syndrome and patients without MS (specificity) | at Baseline
  differentiation between patients with MS and clinically isolated syndrome and patients without MS by analyzing the combination of the presence of CL/LCLs and CVs as compared to the sensitivity/specificity achieved by either CL/LCLs or CVs (sensitivity)
differentiation between patients with MS and clinically isolated syndrome and patients without MS ((specificity) | at Baseline
  differentiation between patients with MS and clinically isolated syndrome and patients without MS by analyzing the combination of the presence of CL/LCLs and CVs as compared to the sensitivity/specificity achieved by either CL/LCLs or CVs (sensitivity)
specificity of the combination of CLs/ LCLs compared to the one of the current diagnostic criteria for MS diagnosis | at Baseline
  specificity of the combination of CLs/ LCLs compared to the one of the current diagnostic criteria for MS diagnosis
sensitivity of the combination of CLs/ LCLs compared to the one of the current diagnostic criteria for MS diagnosis | at Baseline
  sensitivity of the combination of CLs/ LCLs compared to the one of the current diagnostic criteria for MS diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Granziera, Prof., Principal Investigator — Translational Imaging in Neurology, University Hospital Basel
Locations (1):
- Translational Imaging in Neurology, University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Result] La Rosa F, Wynen M, Al-Louzi O, Beck ES, Huelnhagen T, Maggi P, Thiran JP, Kober T, Shinohara RT, Sati P, Reich DS, Granziera C, Absinta M, Bach Cuadra M. Cortical lesions, central vein sign, and paramagnetic rim lesions in multiple sclerosis: Emerging machine learning techniques and future avenues. Neuroimage Clin. 2022;36:103205. doi: 10.1016/j.nicl.2022.103205. Epub 2022 Sep 24. PMID 36201950
- See also: Cortical lesions, central vein sign, and paramagnetic rim lesions in multiple sclerosis: Emerging machine learning techniques and future avenues — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC9668629/